CLINICAL TRIAL: NCT04235634
Title: Evaluation of an Intra-arterial Prostaglandin Therapy in Non-occlusive Mesenteric Ischemia (NOMI)
Brief Title: Intra-arterial Prostaglandin Therapy in Non-occlusive Mesenteric Ischemia
Acronym: REPERFUSE
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: REPERFUSE_8092_BO_S_2018
Record Dates: First submitted 2020-01-13; First posted 2020-01-22 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Non-Occlusive Mesenteric Ischaemia (NOMI)
Keywords: Non-occlusive mesenteric ischemia; Shock; Intra-arterial prostglandin therapy
MeSH Terms: conditions — Shock | interventions — Alprostadil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intra-arterial Prostglandin therapy: Minimal invasive Cannulation of the Superior Mesenteric Artery (SMA) and subsequent intra-arterial application of prostaglandin E1 (Initial Bolus 20ug, followed by continuous Infusion of 60-80ug/24hr for 24-72hrs)
  Interventions: Drug: Prostavasin

INTERVENTIONS:
Drug: Prostavasin — Minimal invasive Cannulation of the Superior Mesenteric Artery (SMA) and subsequent intra-arterial application of prostaglandin E1 (Initial Bolus 20ug, followed by continuous Infusion of 60-80ug/24hr for 24-72hrs)

SUMMARY:
Minimal invasive intra-arterial prostaglandin therapy is currently being offered as an established and safe treatment approach for Non-occlusive mesenteric ischemia (NOMI). So far, there are no data that prospective evaluate clinical response parameters of this method and corresponding criteria for response.

The investigators are therefore planning a prospective observational study on NOMI patients with the aim to collect

1. routine clinical data,
2. data from advanced angigraphic imaging and
3. data from blood biomarkers of intestinal ischemia before/at implementation of intra-arterial vasodilatory therapy.

From these three data packages, the investigators hope to subsequentially derive criteria to better predict response to therapy.

ELIGIBILITY:
Inclusion Criteria:

- persistent shock: Norepinephrine dose > 0.2ug/kg/min over > 48hrs

and

* intestinal failure: paralytic ileus > 24hrs despite neostigmine therapy or
* new onset progressive organ failure (2 out of six criteria): Norepinephrine dose increase, rise in serum lactate, decrease in Horowitz index, new renal replacement therapy, rise in bilirubin, rise in INR, or all of the following: rise in ALT, AST, CK and LDH

Exclusion Criteria:

* patients < 18 years old
* pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with persistent shock, intestinal failure as well as new onset and progressive organ failure with a CT and angiography based diagnosis of Non-occlusive mesenteric ischemia (NOMI)
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Improvement of ischemia | 24 hours following intervention
  Lactate reduction > 2mmol/l from baseline

SECONDARY OUTCOMES:
28-day mortality | 28 days following intervention
  key secondary outcome
Change of norepinephrine dose in microgram/kg/min from baseline at 24 hours | 24 hours following intervention
  as indicator of Shock reversal
simplified NOMI score, range 0-7 points with higher scores indicating more severe NOMI | immediately following first intra-arterial bolus
  angiographic characteristics of vasodilation following Initial Prostaglandin bolus
peak density (PD) as measured by 2D perfusion angiography | immediately following first intra-arterial bolus
  angiographic characteristics of vasodilation following Initial Prostaglandin bolus
area under the curve (AUC) as measured by 2D perfusion angiography | immediately following first intra-arterial bolus
  angiographic characteristics of vasodilation following Initial Prostaglandin bolus
time to peak (TTP) as measured by 2D perfusion angiography | immediately following first intra-arterial bolus
  angiographic characteristics of vasodilation following Initial Prostaglandin bolus
intestinal fatty acid-binding protein (I-FABP), smooth muscle protein of 22kDa (SM22) liver fatty acid-binding protein (L-FABP) | 24 hours following intervention
  markers of ischemic intestinal barrier dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Markus Busch, MD, Principal Investigator — Clinic for gastroenterology and hepatology; Klaus Stahl, MD, Principal Investigator — Clinic for nephrology
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rittgerodt N, Pape T, Busch M, Becker LS, Schneider A, Wedemeyer H, Seeliger B, Schmidt J, Hunkemoller AM, Fuge J, Knitsch W, Fegbeutel C, Gillmann HJ, Meyer BC, Hoeper MM, Hinrichs JB, David S, Stahl K. Predictors of response to intra-arterial vasodilatory therapy of non-occlusive mesenteric ischemia in patients with severe shock: results from a prospective observational study. Crit Care. 2022 Apr 4;26(1):92. doi: 10.1186/s13054-022-03962-w. PMID 35379286